CLINICAL TRIAL: NCT04610658
Title: Activity and Enhancement of Immune Checkpoint Inhibition With Lurbinectedin in Relapsed/Recurrent Small Cell Lung Cancer (SCLC)
Brief Title: Immune Checkpoint Inhibition With Lurbinectedin Relapsed/Recurrent SCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: DLTs
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry); Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20332
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Small-cell Lung Cancer; Relapsed Small Cell Lung Cancer; Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Nivolumab; Ipilimumab; PM 01183

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 Dose Level 1: Nivolumab and Ipilimumab plus Lurbinectedin (Experimental): Participants will be treated at dose level 1: nivolumab 1mg/kg, ipilimumab 3mg/kg plus 1.5 mg/m^2 lurbinectedin. Participants will receive nivolumab, ipilimumab and Lurbinectedin every 3 weeks for 4 cycles. After 4 treatment cycles, ipilimumab will be discontinued and participants will continue treatment with a flat dose of 360 mg nivolumab and Lurbinectedin at dose level 1 every 3 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Lurbinectedin
- Phase 1 Dose Level 2: Nivolumab and Ipilimumab plus Lurbinectedin (Experimental): Participants will be treated at dose level 2: nivolumab 1mg/kg, ipilimumab 3mg/kg plus 2.6 mg/m^2 lurbinectedin. Participants will receive nivolumab, ipilimumab and Lurbinectedin every 3 weeks for 4 cycles. After 4 treatment cycles, ipilimumab will be discontinued and participants will continue treatment with a flat dose of 360 mg nivolumab and Lurbinectedin at dose level 2 every 3 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Lurbinectedin
- Phase 1 Dose Level 3: Nivolumab and Ipilimumab plus Lurbinectedin (Experimental): Participants will be treated at dose level 3: nivolumab 1mg/kg, ipilimumab 3mg/kg plus 3.2 mg/m^2 lurbinectedin. Participants will receive nivolumab, ipilimumab and Lurbinectedin every 3 weeks for 4 cycles. After 4 treatment cycles, ipilimumab will be discontinued and participants will continue treatment with a flat dose of 360 mg nivolumab and Lurbinectedin at dose level 3 every 3 weeks.
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: Lurbinectedin

INTERVENTIONS:
Drug: Nivolumab — Participants will receive 1 mg/kg Nivolumab on Day 1 of each treatment cycle for 4 cycles (induction immunotherapy). After 4 treatment cycles, Nivolumab will be continued at a flat dose of 360 mg.
  Other Names: Opdivo
Drug: Ipilimumab — Participants will receive 3mg/kg Ipilimumab on Day 1 of each treatment cycle for 4 cycles (induction immunotherapy). After 4 cycles, Ipilimumab will be discontinued.
  Other Names: Yervoy
Drug: Lurbinectedin — Participants will be treated at 1 of 3 dose levels of Lurbinectedin, beginning at 1.5 mg/m^2 and increasing to 3.2 mg/m^2 or the Maximum Tolerated Dose (MTD)

SUMMARY:
This is a single-arm, phase I/II trial to determine the Maximum Tolerated Dose (MTD), Recommended Phase II Dose (RP2D), and the safety and efficacy of the combination of nivolumab-ipilimumab plus lurbinectedin in patients with relapsed/recurrent small cell lung cancer after progression with first-line, platinum-based chemotherapy

DETAILED DESCRIPTION:
Study was originally designed as a Phase I/II but was terminated during the Phase I portion due to dose limiting toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Measurable disease based on RECIST v1.1
* Performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Adequate organ function as defined per protocol
* Women of child bearing potential (WOCBP) must have a negative urine or serum pregnancy test within 72 hours from receiving first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* WOCBP should agree to use 2 methods of birth control or abstain from heterosexual activity for the course of the study through 5 months after the last dose of study medication, or should be surgically sterile. Note: A woman is considered to be of "reproductive potential" (WOCBP) if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures, she is responsible for beginning contraceptive measures.
* Male participants should agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy.

Note: In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (vasectomy). However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures, he is responsible for beginning contraceptive measures.

Exclusion Criteria:

Individuals meeting any of the following criteria will be excluded from participation in this study:

* Is currently participating in a study of an investigational agent or device and received or used the investigational agent or device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid or any other form of immunosuppressive therapy within 7 days prior to the first dose of treatment. Note: Systemic steroid doses of ≤ 10 mg of prednisone daily or its equivalent are allowed in patients receiving physiologic replacement steroid doses
* Has a known history of active Bacillus Tuberculosis (TB)
* Hypersensitivity to Lurbinectedin, Ipilimumab and/or nivolumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had targeted small molecule therapy, or standard fractionated radiotherapy within 2 weeks, chemotherapy within 3 weeks and stereotactic radiotherapy within 1 week prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent. Note:: Participants with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study. If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. Other malignancies that remain without evidence of disease or recurrence, 2 years or more after curative therapy are also considered part of this exception.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 2 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has any of the following concomitant diseases/conditions:

  1. History or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically significant valvular heart disease within last year.
  2. Symptomatic arrhythmia or any uncontrolled arrhythmia requiring ongoing treatment.
  3. History of idiopathic, pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis or evidence of active pneumonitis on screening chest CT-scan. History of radiation pneumonitis in radiation field (fibrosis) is permitted, as long as it is asymptomatic and no steroids are needed.
  4. Myopathy or any clinical situation that causes significant and persistent elevation of CPK (>2.5 x upper limit of normal (ULN) in two different determinations performed one week apart).
* Any diagnosis of autoimmune disease (confirmed by medical records or appropriate laboratory testing) is not allowed.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Patients who had a prior Grade ≥3 immune-related adverse event (e.g. pneumonitis, hepatitis, colitis, endocrinopathy) with prior immunotherapy (e.g. cancer vaccine, cytokine, etc.).
* Patients must not be pregnant or nursing due to risk of fetal or nursing infant harm. WOCBP must have agreed to use an effective contraceptive method.
* Participants with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity.
* Participants who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Phase 1: Maximum Tolerated Dose (MTD) of Lurbinectedin with Nivolumab and Ipilimumab | Up to 12 weeks per cohort
  Maximum tolerated Dose will be determined by testing increasing doses of Lurbinectedin along with fixed doses of Nivolumab and Ipilimumab.
Phase II: Disease Control Rate | Up to 12 months
  Disease Control Rate (DCR) is defined as Complete Response (CR) +Partial Response (PR) +Stable Disease (SD). Best response time will be used for this measurement.

SECONDARY OUTCOMES:
Overall Response Rate | Up to 12 months
  Overall Response Rate is defined as Complete Response + Partial Response using RECIST v1.1 criteria.
Progression Free Survival | Up to 12 months
  Progression Free Survival is defined as the time from enrollment to date of progression or death, or censor at last clinical follow-up date.
Overall Survival | Up to 12 months
  Overall Survival is defined as the time from study enrollment to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto A Chiappori, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Advent Health - Celebration, Kissimmee, Florida
  - Moffitt Cancer Center, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Undecided